CLINICAL TRIAL: NCT00653523
Title: Open-label, Long-term Study of Coadministration of Ezetimibe and Simvastatin in Patients With Primary Hypercholesterolemia Who Have Not Reached LDL-cholesterol Target With HMG-CoA Reductase Inhibitors
Brief Title: Coadministration of Ezetimibe and Simvastatin in Patients With Primary Hypercholesterolemia (P05457)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: P05457
Record Dates: First submitted 2008-04-01; First posted 2008-04-07 (Estimated); Results first posted 2010-06-30 (Estimated); Last update posted 2024-05-21 (Actual); Status verified 2022-02

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Ezetimibe; Simvastatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Ezetimibe + Simvastatin (Experimental): Ezetimibe 10 mg + Simvastatin 20 mg
  Interventions: Drug: Ezetimibe; Drug: Simvastatin

INTERVENTIONS:
Drug: Ezetimibe — Ezetimibe 10 mg once daily
  Other Names: SCH 58235
Drug: Simvastatin — Simvastatin 20 mg daily

SUMMARY:
Evaluate the safety of the long-term (1 year) coadministration of ezetimibe and simvastatin in patients with hypercholesterolemia who have not reached low density lipoprotein (LDL)-cholesterol target with 3-hydroxy-3-methylglutaryl coenzyme A (HMG-CoA) reductase inhibitors.

ELIGIBILITY:
Inclusion Criteria:

* Patients with hypercholesterolemia who satisfy the following criteria:

  * Patients who have used any of the following HMG-CoA reductase inhibitors (hereinafter referred to as "statins") for 4 weeks or longer before the start of the observation period and whose LDL-cholesterol level during the treatment had not reached lipid management target indicated below
  * Age: 20 years of age or older (at the time of obtaining informed consent)
  * Sex: both males and females
  * Inpatient/outpatient: Out-patients

Exclusion Criteria:

* Patients for whom any of the following is applicable:

  * Patients whose fasted triglyceride level measured at the start of the observation period or the treatment period exceeds 500 mg/dL
  * Patients with homozygous familial hypercholesterolemia
  * Patients with creatine phosphokinase (CPK) > 2x upper limit of normal (ULN) measured at the start of the observation period or the treatment period.
  * Patients with serious hepatic disorder, or patients with alanine aminotransferase (ALT) or aspartate aminotransferase (AST) > 2x ULN measured at the start of the observation period or the treatment period.
  * Patients with a history of hypersensitivity to any ingredient of ezetimibe tablets or simvastatin tablets
  * Pregnant, nursing women, women who may be pregnant, or patients wishing to be pregnant during the study.
  * Patients who have discontinued use of serum lipid lowering agents for less than 4 weeks at the start of the treatment period (8 weeks in the case of probucol). (However, if the patient had taken a serum lipid lowering agent before the test conducted at the start of the observation period, a period of discontinuation of 27 days, or 55 days in the case of probucol, is allowed.)
  * Patients who are using cyclosporine from after the start of the observation period
  * Patients who are using any of the following drug from after the start of the observation period: itraconazole, miconazole, atazanavir, saquinavir mesilate
  * Patients with a history of ezetimibe use
  * Patients with hyperlipidemia associated with the following diseases:

    * Hypothyroidism
    * Obstructive gall bladder or biliary disease
    * Chronic renal failure
    * Pancreatitis
  * Patients with hyperlipidemia associated with concomitant use of drugs having adverse effect on serum lipids, etc
  * Patients who have received an investigational drug within 4 weeks of the start of the observation period
  * Other patients deemed not appropriate for study entry by the investigator

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2007-12-01 (Actual); Primary Completion 2009-06-01 (Actual); Study Completion 2009-06-01 (Actual)

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Ezetimibe + Simvastatin: Ezetimibe 10 mg + Simvastatin 20 mg
  1. level below what was specified in inclusion criterion
  2. level >2x upper limit of normal at start of treatment
  3. level >=3x upper limit of normal after start of treatment
  4. did not resolve or improve after dose reduction of simvastatin
Period: Overall Study
Arm/Group | Ezetimibe + Simvastatin
Started | 151
Completed | 132
Not Completed | 19
Not completed — Drop in low density lipoprotein (1) | 2
Not completed — Elevated creatine phosphokinase (2) | 1
Not completed — Adverse Event | 7
Not completed — Withdrawal by Subject | 6
Not completed — Elevated alanine aminotransferase (3) | 2
Not completed — Adverse reaction did not improve (4) | 1

BASELINE CHARACTERISTICS:
Arm/Group | Ezetimibe + Simvastatin
Number analyzed (Participants) | 151
Age, Customized [Number; unit: Participants] — Age 20 years and older
  Participants | 151
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82
  Male | 69
Region of Enrollment [Number; unit: participants]
  Japan | 151

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Adverse Events and Adverse Reactions
Description: An adverse event is any unfavorable medical event occurring in a subject to whom an investigational product is administered, and a causal relationship between the administered investigational product and an adverse event is not always clarified.
  That is, an adverse event is any unfavorable or unintended sign (including an abnormal change in laboratory test values), symptom, or disease, and a causal relationship to the relevant investigational product is not considered.
  Any adverse event that was treatment-related was considered an adverse reaction.
Time Frame: Throughout 1 year of study
Measure: Number; unit: Participants
Arm/Group | Ezetimibe + Simvastatin
Number analyzed (Participants) | 151
Participants
  Adverse Events | 143
  Adverse Reactions | 36

ADVERSE EVENTS:
Arm/Group | Ezetimibe+Simvastatin
Serious Adverse Events (participants affected / at risk) | 17/151
Other Adverse Events (participants affected / at risk) | 127/151
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe+Simvastatin (N=151)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 1 (1)
ANGINA UNSTABLE (Cardiac disorders) | 1 (1)
HYPERTROPHIC CARDIOMYOPATHY (Cardiac disorders) | 1 (1)
EYE PAIN (Eye disorders) | 1 (1)
PNEUMONIA (Infections and infestations) | 1 (1)
CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 3 (3)
IN-STENT CORONARY ARTERY RESTENOSIS (Injury, poisoning and procedural complications) | 1 (2)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 1 (1)
ROTATOR CUFF SYNDROME (Musculoskeletal and connective tissue disorders) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
UTERINE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
SUBARACHNOID HAEMORRHAGE (Nervous system disorders) | 1 (1)
ACTINIC KERATOSIS (Skin and subcutaneous tissue disorders) | 1 (1)
ARTERIAL STENT INSERTION (Surgical and medical procedures) | 1 (2)
AORTIC DISSECTION (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ezetimibe+Simvastatin (N=151)
CONSTIPATION (Gastrointestinal disorders) | 9 (9)
BRONCHITIS (Infections and infestations) | 20 (25)
NASOPHARYNGITIS (Infections and infestations) | 46 (73)
PHARYNGITIS (Infections and infestations) | 10 (13)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 26 (32)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 10 (11)
BLOOD AMYLASE INCREASED (Investigations) | 12 (14)
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 27 (33)
C-REACTIVE PROTEIN INCREASED (Investigations) | 41 (47)
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 14 (14)
GLYCOSYLATED HAEMOGLOBIN INCREASED (Investigations) | 10 (11)
MYOGLOBIN BLOOD INCREASED (Investigations) | 21 (21)
WHITE BLOOD CELL COUNT INCREASED (Investigations) | 12 (12)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 8 (8)
HYPOGLYCAEMIA (Metabolism and nutrition disorders) | 9 (14)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 15 (15)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 17 (17)
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 14 (20)
MUSCULOSKELETAL STIFFNESS (Musculoskeletal and connective tissue disorders) | 13 (14)
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 11 (12)
HEADACHE (Nervous system disorders) | 12 (14)
UPPER RESPIRATORY TRACT INFLAMMATION (Respiratory, thoracic and mediastinal disorders) | 11 (13)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Principal Investigator (PI) agrees, for a period of 5 years following the Effective Date, to retain the Disclosure made to it by or on behalf of Sponsor (SPKK), in confidence and not to disclose it to any third party.

PI further agrees that during such time period it will not, either directly or indirectly, use the Disclosure for any purpose(s) other than that indicated herein without the prior written consent of SPKK.